CLINICAL TRIAL: NCT00273338
Title: A Phase 3, Randomized, Open-Label Study Evaluating DN-101 in Combination With Docetaxel in Androgen-Independent Prostate Cancer (AIPC) (ASCENT-2)
Brief Title: DN-101 in Combination With Docetaxel in Androgen-Independent Prostate Cancer (AIPC) (AIPC Study of Calcitriol Enhancing Taxotere [ASCENT-2])
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB
Sponsor: Novacea (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011-007
Record Dates: First submitted 2005-12-14; First posted 2006-01-09 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer
Keywords: Androgen-independent Prostate Cancer (AIPC); Prostate Cancer; DN-101; calcitriol; Taxotere; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Docetaxel

INTERVENTIONS:
Drug: calcitriol
Drug: docetaxel

SUMMARY:
The primary objective of this study is:

* To evaluate the effect of DN-101 in combination with docetaxel (ASCENT regimen) on survival in metastatic androgen-independent prostate cancer

The secondary objectives of this study are:

* To determine the effect of the ASCENT regimen on the rate of thromboembolic events (blood clots)
* To determine the effect of the ASCENT regimen on prevention of skeletal-related events (fractures)
* A Separate sub-study will be conducted at selected study sites in North America to determine the population PK of DN-101.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically proven adenocarcinoma of the prostate
* Documented metastatic prostate adenocarcinoma
* Documented progression while on androgen ablation therapy detected by rising prostate specific antigen (PSA) and/or imaging
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* Adequate hematologic, renal and hepatic function
* Life expectancy >= 3 months

Exclusion Criteria:

* Prior chemotherapy, except estramustine
* Prior chemotherapy with docetaxel
* Prior isotope therapy (e.g., strontium-89, samarium-153, etc.)
* One or more contraindications to the use of corticosteroids
* History of cancer-related hypercalcemia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard I. Scher, MD, Study Chair — Sidney Kimmel Center for Prostate and Urologic Cancers, Memorial Sloan Kettering Cancer Center; Kim N. Chi, M.D., Study Chair — British Columbia Cancer Agency - Vancouver Centre; Ronald De-Wit, M.D., Study Chair — Erasmus University Medical Center (Netherlands)
Locations (222):
- United States (159):
  - Birmingham Hematology & Oncology Associates, LLC, Birmingham, Alabama
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Hematology Associates - AOA, Phoenix, Arizona
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Northern Arizona Hematology & Oncology Associates, AOA, Sedona, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - U of Arizona / Arizona Cancer Center, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Pacific Shores Medical Group, Long Beach, California
  - The Angeles Clinic and Research Institute, Inc., Los Angeles, California
  - UCLA department of Urology, Los Angeles, California
  - Veterans Affairs Northern California Health Care System, Martinez, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Monterey Bay Oncology, Monterey, California
  - Comprehensive Cancer Center at, Palm Springs, California
  - Sutter Cancer Center, Sacramento, California
  - UCD Cancer Center-Clinical Trials, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Georgetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - Pasco Hernando Oncology Associates, P.A., 14529 Cortez Blvd., Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, U of Miami, Miami, Florida
  - Pasco Hernando Oncology Associates P.A., New Port Richey, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Innovative Medical Research of South Florida Inc., North Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - AYS Urology, Trinity, Florida
  - Phoebe Cancer Center, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Peachtree Hematology-Oncology Consultants, PC, Atlanta, Georgia
  - Atlanta Cancer Care, Atlanta, Georgia
  - Northeast GA Medical Center, Gainesville, Georgia
  - Georgia Cancer Specialist, Tucker, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Midwest Prostate & Urology Health Center, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - Swedish American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates of Illinois, L.L.C, Skokie, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Medical Consultants, PC c/o Ball Cancer Center, Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Hope Center, Terre Haute, Indiana
  - Medical Center of Vincennes, Vincennes, Indiana
  - Iowa Cancer Care, Cedar Rapids, Iowa
  - Mercy Medical Center, North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - St. Agnes Health System, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - MN Cooperative Group Outreach Prg., Minneapolis, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - University of Missouri, Ellis Fischel Cancer Center, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Nebraska Methodist Hospital - Oncology Research Dept, Omaha, Nebraska
  - Horizon's West Medical Group, Scottsbluff, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - UMDNJ-Newark, Newark, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Overlook Oncology Center, Summit, New Jersey
  - New Mexico Cancer Care Associates, Sante Fe, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Hematology Oncology Associates of, New City, New York
  - Memorial Sloan-Kett, New York, New York
  - Interlakes Foundation Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Staten Island Urological Research, PC, Staten Island, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Carolina Cancer Management, Inc., Fayetteville, North Carolina
  - Piedmont Hematology Oncology Associates, PLLC, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Mid Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Dayton Oncology & Hematology, P.A., Kettering, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Consultants in Medical Oncology & Hematology, Drexel Hill, Pennsylvania
  - Hematology & Oncology Associates of Northeastern PA, Dunmore, Pennsylvania
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Greater Philadelphia Cancer, Philadelphia, Pennsylvania
  - Univeristy of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottsville Cancer Care, Pottsville, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Charleston Hematology Oncology PA, Charleston, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolina, Greenville, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Chattanooga Oncology & Hematology Assoc., Chattanooga, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Cancer Center-Abilene, Abilene, Texas
  - Texas Oncology, PA, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Urology Associates of North Texas (UANT), Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - MamieMcFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Cancer Center ar Medical City, Dallas, Texas
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Center-East, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - The Center for Cancer & Blood Disorders, Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Texas Oncology, P.A., Longview, Texas
  - Southwest Cancer Treatment and Research Center, Lubbock, Texas
  - South Texas Cancer Center - McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - Cancer Care Network of South Texas, HOAST, New Braunfels, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - South Texas Oncology and Hematology, PA, San Antonio, Texas
  - InVisions Consultants LLC, San Antonio, Texas
  - Texas Cancer Center- Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Texas Oncology, Waco, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Fairfax Northern Virginia Hematology OnCology, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Centers, Edmonds, Washington
  - University of Washington, Seattle, Washington
  - Puget Sound Cancer Centers, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (18):
  - Tom Baker Cancer Center-Medical Oncology, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital (SERHA), Moncton, New Brunswick
  - Dr. Leon Richard Oncology Center, Moncton, New Brunswick
  - Centre for Clinical Research Cancer Care Program, Halifax, Nova Scotia
  - Regional Cancer Program de l'Hopital Regional de Sudbury, Greater Sudbury, Ontario
  - Jaravinski Cancer Centre Hamilton Health Services, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - McGill University, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Czechia (3):
  - Institute of Radiation Oncology of Teaching Hospital Na Bulovce, Prague
  - Department of Radiation and Oncology of Teaching Hospital Motol, Prague
  - Teaching Hospital Kralovske Vinohrady, Prague
- Germany (28):
  - Universitätsklinikum Köln, Cologne, 50931
  - Gemeinschaftspraxis für Hämatologie & Onkologie, Augsburg
  - Facharzt f. Urologie, Bad Schwartau
  - Urologische Praxis, Bautzen
  - Universitatsmedizin Charité, Berlin
  - Klinik am Urban, Berlin
  - Universitätsmedizin Charité Campus Benjamin Franklin, Berlin
  - Urologische Praxis, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Facharzt f. Urologie, Cottbus
  - Urologische Klinik, Dresden
  - Universitäsklinikum Düsseldorf, Düsseldorf
  - Urologische Klinik der Universitätsklink Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum Fulda, Urologische Klinik, Fulda
  - Urologische Praxis, Hagenow
  - Urologische Gemeinschaftspraxis, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum Homburg/Saar, Homburg
  - Klinikum Kassel GmbH, Kassel
  - Gemeinschaftspraxis für Urologie, Kirchheim/Teck
  - Gesellschaft f. klinische Studien und Urologisches Gesundheitszentrum, Leipzig
  - Oberarzt d. Urolog. Abteilung, München
  - Obearzt der Urologischen Klinik, Universitätsklinik Münster, Münster
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - Gemeinschaftspraxis f. Urologie, Wuppertal
  - Urologische Praxis, Zwickau
- Hungary (4):
  - IRM Center Hospital and Institutes, II.Department of Oncology, Budapest
  - Uzsoki Hospital of the Local Authority of Budapest, Oncoradiology, Budapest
  - University of Debrecen, Medical and Health Science Center, Department of Oncology, Debrecen
  - University of Szeged, Szent-Györgyi Albert Medical and Pharmacist Science Center, Clinic of Oncotherapy, Szeged
- San Juan VA Medical Center, Reseach Dept, San Juan, Puerto Rico
- Romania (5):
  - Cabinetul de Urologie, Arad
  - Policlinica de diagnostic rapid, Brasov
  - Institutul Oncologic Bucuresti, Bucharest
  - Euro S.R.L., Cluj-Napoca
  - ProVita 2000, Constanța
- Clinical Center Niš - Clinic of Urology, Belgrade, Serbia and Montenegro
- Slovakia (3):
  - Theaching Hospital of F.D. Roosevelt, Banská Bystrica
  - Faculty Hospital Martin, Martin
  - Faculty Hospital of J. A. Reiman, Prešov